CLINICAL TRIAL: NCT06802744
Title: Changes in Systemic Carbon Dioxide Levels During Simulated Avalanche Burial Using a One-way Valve Device: a Double Blinded, Randomized Cross-over Trial
Brief Title: Changes in the Carbon Dioxide Content in the Body During a Simulated Avalanche Burial With and Without the Use of a Breathing Tube System.
Acronym: Avalanox
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Klinik fur Pneumologie und Schlafmedizin Kantonsspital Aarau (Industry)
Responsible Party: Principal Investigator, Hans-Joachim Kabitz, Prof. Dr. med., Kantonsspital Aarau
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2024-02335
Record Dates: First submitted 2025-01-20; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Avalanche Burial
Keywords: AAPD; Artificial air-pocket device

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulated avalanche burial using a artificial air-pocket device (Experimental)
  Interventions: Device: Addition of an artificial air-pocket device during simulated avalanche burial
- Simulated avalanche burial using a non-functional artificial air-pocket device (Sham Comparator)
  Interventions: Device: Addition of a non-functioning artificial air-pocket device during simulated avalanche burial

INTERVENTIONS:
Device: Addition of an artificial air-pocket device during simulated avalanche burial — In contrast to the control group, the subjects in this arm are provided with a functioning device that directs the exhaled air away from the area of the respiratory cavity.
  Arms: Simulated avalanche burial using a artificial air-pocket device
Device: Addition of a non-functioning artificial air-pocket device during simulated avalanche burial — In contrast to the intervention arm, the subjects in this arm are provided with a non-functioning artificial air-pocket device which does not redirect the exhaled air away from the breathing-cavity.
  Arms: Simulated avalanche burial using a non-functional artificial air-pocket device

SUMMARY:
Every year, around 100 people die in avalanches in the Alps. Many of these accidents occur during winter sports. In most cases, the victims suffocate under the snow after the avalanche has come to a standstill. A key survival factor here is the time it takes to be rescued. If a buried victim is rescued within 15 minutes, the probability of survival is over 90%. After 35 minutes, however, this drops drastically to just 30%.

A modern avalanche rescue system, such as the AvaLung-device, could extend the survival time. The system directs the exhaled air via a tube to the back of the buried person so that no toxic CO2 concentrations build up in the available breathing cavity. It is also intended to prevent the formation of an "ice mask", which can impair the release of oxygen from the snow. This study investigates whether the AvaLung system can extend the survival time in the event of burial.

The aim is to test the effects of such a breathing tube system. The oxygen and carbon dioxide levels of the test subjects are measured while they are buried in a simulated avalanche - once with and once without the AvaLung system. In addition, it is investigated how long it takes before the buried subjects have to stop the examination, for example due to shortness of breath or deteriorating respiratory gases in the blood.

Test setup:

The test subjects lie on their backs with their heads and chests buried under snow. During the test phase, various parameters are continuously monitored, such as the breathing rate and the CO2 concentration in the blood. A comparative study is carried out: once with a functioning rescue system, and once with a manipulated (non-functioning) system.

Expected benefit:

The results of this study should contribute to a better understanding of the effectiveness of avalanche rescue systems and thus increase the chances of survival of avalanche victims in the future. This is particularly important today, as the number of winter sports enthusiasts and the number of avalanches triggered by them is constantly increasing.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18
* Able to consent

Exclusion Criteria:

* Anamnestic evidence of previous pulmonary or cardiac disease
* Known neuromuscular diseases
* Thoracic deformities
* Acute respiratory infections
* In women: Pregnancy (excluded by history and urine test)
* Age over 60 Years
* Presence of claustrophobia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-07 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Course of PtCO2 measured transcutaneously | 45 minutes

SECONDARY OUTCOMES:
Burial time until the test is terminated | 45 minutes
Course of PetCO2 | 45 minutes
Progression of respiratory minute volume | 45 minutes
Course of the body temperature | 45 minutes
Heart rate progression and variability | 45 minutes
Course of PtO2 | 45 minutes
Course of PetO2 | 45 minutes
Course of SpO2 | 45 minutes
Progression of Respiratory rate | 45 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Joachim Kabitz, Prof. Dr. med., Principal Investigator — Klinik für Pneumologie und Schlafmedizin Kantonsspital Aarau
Locations (1):
- Kantonsspital Aarau, Aarau, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided